CLINICAL TRIAL: NCT03859908
Title: Iodine-Povidone Alcohol Compared to Chlorhexidine Alcohol as Preoperative Antiseptics in Major Abdominal Elective Clean Contaminated Surgery
Brief Title: Comparison of Two Preoperative Antiseptic Solutions Alcohol Based in Abdominal Elective Surgeries
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties for recruitment due to COVID-19 pandemia and expiration of the material
Sponsor: Universidad de El Salvador (Other)
Responsible Party: Principal Investigator, Maria-Virginia Rodriguez Funes, Clinical research coordinator, Universidad de El Salvador
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Iodine alcohol Trial; CNEIS/2018/049 (Other: Comite Nacional de Etica de Investigacion en Salud)
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Surgical Site Infection
Keywords: surgery; infection; antisepsis
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — 2-Propanol; DuraPrep; chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Pragmatic, randomized controlled trial of two substances
Who Masked: Participant
Masking Description: Participant will be randomized through a selection of a sealed envelope with computer generated random numbers by the Operating Room nurse, and the substance will be applied when participant will be already with anesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Iodine-Povacrylex Alcohol (Experimental): Iodine Povacrylex 7 MG/ML / Isopropyl Alcohol 0.74 ML/ML: preoperative asepsis with subject already lying down in the operating room, already with anesthesia, before dressing and incision, with single dose applicator of Iodine-povacrylex 7mg/ml plus isopropyl alcohol 0.74 ml/ml (DuraPrep) , fabricated by 3M, as the experimental intervention. Will be applied from the center of the abdomen centrifuge as recommended by the Centers of Disease Control
  Interventions: Drug: Iodine Povacrylex 7 MG/ML / Isopropyl Alcohol 0.74 ML/ML
- Chlorhexidine Alcohol (Active Comparator): Chlorhexidine Gluconate 20 MG/ML / Isopropyl Alcohol 0.7 ML/ML: preoperative asepsis with subject already lying down in the operating room, already with anesthesia, before dressing and incision, with single dose applicator of chlorhexidine 20 mg/ml plus isopropyl alcohol 0.7 ml/ml (SoluPrep), fabricated by 3M, as the control intervention. Will be applied from the center of the abdomen centrifuge as recommended by the Center of Disease Control
  Interventions: Drug: Chlorhexidine Gluconate 20 MG/ML / Isopropyl Alcohol 0.7 ML/ML

INTERVENTIONS:
Drug: Iodine Povacrylex 7 MG/ML / Isopropyl Alcohol 0.74 ML/ML — As preoperative antiseptic, applied once as suggested by Centers for Disease Control recommendations in surgical asepsis
  Other Names: [DuraPrep]
  Arms: Iodine-Povacrylex Alcohol
Drug: Chlorhexidine Gluconate 20 MG/ML / Isopropyl Alcohol 0.7 ML/ML — As preoperative antiseptic, applied once as suggested by Centers for Disease Control recommendations in surgical asepsis
  Other Names: SoluPrep; ChloraPrep
  Arms: Chlorhexidine Alcohol

SUMMARY:
Pragmatic randomized clinical trial comparing Iodine Povacrylex based on alcohol to Chlorhexidine also based on alcohol in efficacy and security to diminish frequency of surgical site infections in major abdominal elective clean contaminated wounds. Will be held in a third level university, high volume national public hospital in San Salvador, El Salvador.

DETAILED DESCRIPTION:
Preoperative antiseptic Chlorhexidine based on alcohol has been established as gold standard of care for clean contaminated wounds. It was compared to Iodine solutions non-alcohol based. There is a question about alcohol based solution was a confounder in the comparison. The aim of this study is to compare the efficacy of both solutions alcohol based, 0.7% iodine povacrylex plus 74% alcohol, against gluconate chlorhexidine 2% plus 70% alcohol, in clean contaminated wounds, in major abdominal elective surgeries, in a wider range than colorectal surgeries, Materials and methods. With a pragmatic randomized, phase 4, controlled clinical trial. Comparison of two antiseptic solutions, using manufacturer (3M) sterile appliers' for both products, Food and Drugs Agency approved.

Quality of data will be assured by first training all surgeons and residents besides researchers in the study protocol for protocol compliance in subject identification, randomization moment, and follow up. There is a plan for weekly monitoring of protocol compliance, and monthly data monitoring and auditing from Faculty of Medicine Research Unit.

Monitoring and auditing will comply protocol compliance and data integrity against subject's medical records and random interviews of patients in their post-surgical control.

Surgical Site Infection definitions are those taken from Centers for Disease Control definitions.

Standard Operating Procedures will be established in all moments of the trial, from subject identification, informed consent, recruitment, randomization process in the operating room, and data collection in pre specified files for data collection and data management. Protocol compliance and Standard Operating Procedures compliance will be monitored by Principal Investigator constantly. Report of adverse events will be done in accordance to Salvadoran National ethics committee Standard Operating Procedures as also any other communication such as protocol deviance or amendments. Previous research has not reported adverse events, but we will be expectant to their appearance.

Sample size was calculated for a total of 964 subjects, 482 in each group, using statistics software, were we established a statistic significant level for a bilateral hypothesis of 95% and a power of 80%, based on previous research of comparison of both solutions to get a probability of SSI of 4.2% in Chlorhexidine group against 8.6% in Iodine povacrylex group.

We will establish a strict follow up of patients in the 30 days considered as post-operative time, by enabling the whole public health system to integrate in subjects´, surgical care (primary care) to diminish the probability of missing data.

Data analysis will be done following "intention to treat" analysis principle. Primary outcome will be any kind of Surgical Site Infection, categorical variable, will be analyzed with chi square for a bilateral hypothesis, and also measure the difference with risk ratio and its 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery categorized as clean contaminated surgery Major abdominal

-

Exclusion Criteria:

* American Society of Anesthesia III-IV
* Laparoscopic cholecystectomy
* Inguinal hernias classification I, II
* Obese subjects with Body Mass Index more than 35 or malnourished
* immunocompromised subjects
* neoplasia Preoperative hospital stay more than 7 days allergic to any of the solutions used in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | Date of event occurs within 30 days after any operative procedure (where day 1 = the procedure date)
  infections of the incision or organ or space that occur after surgery.

SECONDARY OUTCOMES:
Superficial surgical site infection | Date of event occurs within 30 days after any operative procedure (where day 1 = the procedure date)
  Infection that occurs after surgery and involves only skin and subcutaneous tissue of the incision
Deep surgical site infection | Date of event occurs within 30 days after any operative procedure (where day 1 = the procedure date)
  Infection that occurs after surgery that involves deep soft tissues of the incision (for example, fascial and muscle layers)
Organ/space SSI | Date of event occurs within 30 days after any operative procedure (where day 1 = the procedure date)
  Infection that occurs after surgery that involves any part of the body deeper than the fascial/muscle layers that is opened or manipulated during the operative procedure
Skin reaction | Date of event occurs within 7 days after surgery (where day 1= the procedure date
  Any kind of irritation or skin reaction after applying the solution

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Virginia Rodriguez, MD, FACS, Principal Investigator — Universidad de El Salvador
Locations (1):
- Hospital Nacional Rosales, San Salvador, El Salvador

IPD SHARING:
Plan to Share IPD: No
If we decide to share IPD, it will be: study protocol, statistical analysis. Criteria to share: for systematic reviews we could share also individual data collected, after the study is published.
  The study was stopped for recruitment due to COVID-19 emergency and elective surgeries diminished, and then the product used expired. Couldn't achieve not even 2% of Sample size